CLINICAL TRIAL: NCT03536650
Title: Evaluation of Duodenal Mucosal Resurfacing (DMR) for the Treatment of Non Alcoholic Steatohepatitis (NASH), a Proof of Concept Study
Brief Title: Effect of DMR in the Treatment of NASH
Acronym: DMR_NASH_001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Fractyl Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2017/302
Record Dates: First submitted 2018-04-13; First posted 2018-05-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Metabolic diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DMR procedure (Experimental)
  Interventions: Device: DMR

INTERVENTIONS:
Device: DMR — Procedure: DMR Procedure The Fractyl DMR procedure using the Revita System utilizes an over the wire endoscopic approach to ablate the duodenum. The procedure may be completed in an endoscopic suite or in an operating room depending on the facilities and support at each investigative site. All subjects are monitored and anesthetized by conscious sedation per each facility's standard protocol. A full DMR procedure is defined as 5 complete ablations or 9 axial centimeters of circumferentially ablated tissue in the duodenum. Subjects who do not receive any ablations during the DMR procedure will be followed for safety through the 4 week visit and then discontinued from the study.
  Other Names:
  DMR Revita
  Other Names: Revita

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a frequent disease affecting up to 25% of the USA population, 2-44% in Europe and up to 42,6-69,5% in patients with type 2 diabetes. It is a disease that could progress from simple steatosis to non-alcoholic steatohepatitis (NASH), hepatic cirrhosis and hepatocarcinoma. NASH is part of continuum of metabolic syndrome and constitutes a serious public health concern manifesting by premature cardiovascular disease, end stage diabetes complication and will likely become the first cause of end stage liver disease. Insuline resistance is the hallmark of NASH. Some recent studies both in animals and humans have demonstrated abnormal hypertrophy of the duodenal mucosa, changes in enteroendocrine cell density and number, endocrine hyperplasia, and alterations in gut hormone signaling highlighting the role of the upper intestine gut in glucose homeostasis and thus insulin sensitizing. Given these physiological and pathophysiological features, abrasion of duodenal mucosa was assessed both in animals and humans. The investigators reported an improvement in both glucose homeostasis and transaminases levels suggesting possibly an improvement of NASH. Until now, lifestyle medication is the only recognized efficient treatment for fatty liver disease. Unfortunately, only a minority of patients achieve a significant weight loss and lifestyle modifications. The investigators aim to study the duodenal mucosal resurfacing procedure in patients with NASH biopsy proven in a proof of concept study allowing to assess this technique as a potential treatment to NASH.

DETAILED DESCRIPTION:
Introduction

Non-alcoholic fatty liver disease (NAFLD) is a frequent disease affecting up to 25% of the USA population, 2-44% in Europe and up to 42,6-69,5% in patients with type 2 diabetes. It is a disease that could progress from simple steatosis to non-alcoholic steatohepatitis (NASH), hepatic cirrhosis and hepatocarcinoma. NASH is part of continuum of a metabolic syndrome and constitutes a serious public health concern, manifesting by premature cardiovascular disease, end stage diabetes complication and will likely become the first cause of end stage liver disease.

Insulin resistance is the hallmark of NASH. Some recent studies both in animals and humans have demonstrated abnormal hypertrophy of the duodenal mucosa, changes in enteroendocrine cell density and number, endocrine hyperplasia, and alterations in gut hormone signaling highlighting the role of the upper intestine gut in glucose homeostasis and thus insulin sensitizing.

Given these physiological and pathophysiological features, abrasion of duodenal mucosa was assessed both in animals and humans. The investigators reported an improvement in both glucose homeostasis and transaminases levels suggesting possibly an improvement of NASH.

Until now, lifestyle medication is the only recognized efficient treatment for fatty liver disease. Unfortunately, only a minority of patients achieve a significant weight loss and lifestyle modifications.

The investigators aim to study the duodenal mucosal resurfacing procedure in patients with NASH biopsy proven in a proof of concept study allowing to assess this technique as a potential treatment to NASH.

Design of study The study is designed as a single arm, proof of concept, non-randomized, open label trial to be conducted at one investigational site. All patients with biopsy proven NASH will undergo an upper endoscopy to perform a duodenal mucosal resurfacing procedure. Evolution of liver steatosis (assessed by MRI), insulin resistance (assessed by oral glucose tolerance test), liver damage (evaluated by blood tests), liver elastography (assessed by fibroscan, fibrotest), biometric parameters will be performed pre- and post-procedure.

Primary outcome :

- Feasability and safety of duodenal mucosal resurfacing, using Revita ™ duodenal mucosal resurfacing after submucosal injection, in patients with NASH.

Secondary outcomes:

* Evolution of steatosis assessed by MRI 6 months after the procedure.
* Evolution of liver fibrosis (assessed by Fibroscan, Fibrotest, Fibrosis four score (FIB-4) and NAFLD fibrosis score) at 6 and 12 months after the procedure.
* Evolution of liver tests at 6 and 12 months after the procedure.
* Evolution of insulin resistance at 1,3,6 and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (male and female), age 28 to 75 years.
2. NASH histological diagnosis according to the currently accepted definition of both EASL and AASLD, requiring the combined presence of steatosis (any degree> 5%) + lobular inflammation of any degree + liver cell ballooning of any amount, on a liver biopsy performed ≤ 6 months before screening in the study and confirmed by central reading during the periode and (apendix 1)

   1. SAF (steatosis, activity, fibrosis) activity score of 3 or 4 (>2)
   2. SAF steatosis score ≥ 1
   3. SAF fibrosis score < 4
3. No other causes of chronic liver disease and compensated liver disease.
4. If applicable, have a type 2 diabetes with HbA1c <10.0 %
5. BMI (body mass index) ≥ 24 and ≤ 40 kg/m2.
6. Willing to sign an informed consent form.
7. Willing to comply with study requirements

Exclusion Criteria:

1. Evidence of another cause of liver disease.
2. History of sustained alcohol ingestion defined as: daily alcohol consumption > 30 g/day for males and > 20 g/day for females.
3. Previous gastrointestinal surgery such as subjects who have had Billroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions.
4. Known autoimmune disease, including celiac disease, or symptoms of systemic lupus eythematosus, sleroderma or other auto-immune connective tissue disorder.
5. For type 2 diabetes subjects, no current use of insulin or GLP-1 analogues.
6. Type 1 diabetes.
7. Probable insulin production failure defined as fasting C peptide serum < 1 ng/ml.
8. History of acute or chronic pancreatitis.
9. Active malignancy.
10. Persistent anemia defined as Hb < 10 g/dl.
11. Use of anticoagulation therapy which cannot be discontinued for 7 days before and 14 days after the procedure.
12. Use of P2Y12 inhibitors (clopidrogel, prasugrel, ticagrelor) which cannot be discontinued for 14 days before and14 days after the procedure.
13. History of coagulopathy or upper gastro-intestinal bleeding conditions likely to bleed.
14. Taking corticosteroids or drugs which possibly affect gastrointestinal motility or liver.
15. Unable to discontinue NSAIDs (non-steroidal anti- inflammatory drugs) during the treatment up to 4 weeks after procedure.
16. Use of weight loss medications.
17. Presence of liver cirrhosis (defined by histology)
18. Platelet count < 120 x 109/L.
19. Clinical evidence of hepatic decompensation or severe liver impairment as defined by the presence of any of the following abnormalities:
20. Serum albumin < 32 g/L.
21. INR> 1.3.
22. Direct bilirubin> 1.3 mg/L.
23. ALT or AST > 5x ULN.
24. Alkaline Phosphatase > 3x ULN.
25. History of esophageal varices, ascites or hepatic encephalopathy.
26. Splenomegaly.
27. Human immunodeficiency virus.
28. Contraindications to MRI as defined below.

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Safety of duodenal mucosal resurfacing characterized by the incidence of all Adverse Device Effects (ADEs), and subsequent adverse events [ Time Frame: 12 months ] in patients with NASH. | 12 months
  Safety will be characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants.
  Safety evaluations will also be performed to ensure no subsequent adverse events have occurred and to ensure any adverse events during the trial that are considered on-going are stable or have resolved. Safety will be assessed at 1 and 6 months following the intervention.

SECONDARY OUTCOMES:
Change in Magnetic Resonance Fat Fraction (MRFF) from baseline in the following 6 months in DMR subjects. | baseline and 6 months post-procedure
  Magnetic Resonance Fat fraction
Change in NAS score from baseline in the following 12 months in DMR subjects. | baseline and 12 months post-procedure
  Centrally scored histological improvement in NAFLD from baseline to the end of 12 months post-procedure, where improvement is defined as:
  * No worsening in fibrosis; and
  * A decrease in NAFLD Activity Score (NAS) of at least 2 points
Change in Fibrosis-4 Index for Liver Fibrosis (FIB-4) from baseline in the following at 6 months in DMR subjects | baseline and 6 months post-procedure
  Absolute change in Fibrosis-4 Index for Liver Fibrosis (FIB-4) is a fibrosis marker. A score <1.45 has a negative predictive value of over 90% for advanced liver fibrosis. A score of >3.25 has a positive predictive value of 65% for advanced fibrosis with a specificity of 97%.
Change in Fibrosis-4 Index for Liver Fibrosis (FIB-4) from baseline in the following at 12 months in DMR subjects | baseline and 12 months post-procedure
  Absolute change in Fibrosis-4 Index for Liver Fibrosis (FIB-4) is a fibrosis marker. A score <1.45 has a negative predictive value of over 90% for advanced liver fibrosis. A score of >3.25 has a positive predictive value of 65% for advanced fibrosis with a specificity of 97%.
Change in Transient Elastography using Firboscan from baseline in the following at 6 months in DMR subjects | baseline and 6 months post-procedure
  Transient Elastography
Change in Transient Elastography using Firboscan from baseline in the following at 12 months in DMR subjects | baseline and 12 months post-procedure
  Transient Elastography
Change in Magnetic Resonance Fat Fraction (MRFF) from baseline in the following 12 months in DMR subjects. | baseline and 12 months post procedure
  Magnetic Resonance Fat fraction
Change in transaminases levels from baseline in the following 6 months in DMR subjects | baseline and 6 months post-procedure
  Transaminases levels
Change in transaminases levels from baseline in the following 12 months in DMR subjects | baseline and 12 months post-procedure
  Transaminases levels
Change in Insulin resistance measured by oral glucose tolerance test (OGTT) from baseline in the following 6 months in DMR subjects | baseline and 6 months post-procedure
  Insulin resistance as abnormal HOMA IR
Change in Insulin resistance measured by oral glucose tolerance test (OGTT) from baseline in the following 12 months in DMR subjects | baseline and 12 months post procedure
  Insulin resistance as abnormal HOMA IR
Change in stage of fibrosis from baseline in the following 12 months in DMR subjects | baseline and 12 months post-procedure
  Liver histology

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Deviere, PhD, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Jadhav K, Zhang Y. Bile acid receptors in non-alcoholic fatty liver disease. Biochem Pharmacol. 2013 Dec 1;86(11):1517-24. doi: 10.1016/j.bcp.2013.08.015. Epub 2013 Aug 26. PMID 23988487
- [Background] Blachier M, Leleu H, Peck-Radosavljevic M, Valla DC, Roudot-Thoraval F. The burden of liver disease in Europe: a review of available epidemiological data. J Hepatol. 2013 Mar;58(3):593-608. doi: 10.1016/j.jhep.2012.12.005. PMID 23419824
- [Background] Tilg H, Moschen AR. Evolution of inflammation in nonalcoholic fatty liver disease: the multiple parallel hits hypothesis. Hepatology. 2010 Nov;52(5):1836-46. doi: 10.1002/hep.24001. PMID 21038418
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ; American Gastroenterological Association; American Association for the Study of Liver Diseases; American College of Gastroenterologyh. The diagnosis and management of non-alcoholic fatty liver disease: practice guideline by the American Gastroenterological Association, American Association for the Study of Liver Diseases, and American College of Gastroenterology. Gastroenterology. 2012 Jun;142(7):1592-609. doi: 10.1053/j.gastro.2012.04.001. Epub 2012 May 15. No abstract available. PMID 22656328
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Boza C, Riquelme A, Ibanez L, Duarte I, Norero E, Viviani P, Soza A, Fernandez JI, Raddatz A, Guzman S, Arrese M. Predictors of nonalcoholic steatohepatitis (NASH) in obese patients undergoing gastric bypass. Obes Surg. 2005 Sep;15(8):1148-53. doi: 10.1381/0960892055002347. PMID 16197788
- [Background] Higuera-de la Tijera F, Servin-Caamano AI. Pathophysiological mechanisms involved in non-alcoholic steatohepatitis and novel potential therapeutic targets. World J Hepatol. 2015 Jun 8;7(10):1297-301. doi: 10.4254/wjh.v7.i10.1297. PMID 26052375
- [Background] Schneck AS, Anty R, Patouraux S, Bonnafous S, Rousseau D, Lebeaupin C, Bailly-Maitre B, Sans A, Tran A, Gugenheim J, Iannelli A, Gual P. Roux-En Y Gastric Bypass Results in Long-Term Remission of Hepatocyte Apoptosis and Hepatic Histological Features of Non-alcoholic Steatohepatitis. Front Physiol. 2016 Aug 19;7:344. doi: 10.3389/fphys.2016.00344. eCollection 2016. PMID 27594839
- [Background] Hannah WN Jr, Harrison SA. Effect of Weight Loss, Diet, Exercise, and Bariatric Surgery on Nonalcoholic Fatty Liver Disease. Clin Liver Dis. 2016 May;20(2):339-50. doi: 10.1016/j.cld.2015.10.008. Epub 2016 Feb 17. PMID 27063273
- [Background] Klebanoff MJ, Corey KE, Chhatwal J, Kaplan LM, Chung RT, Hur C. Bariatric surgery for nonalcoholic steatohepatitis: A clinical and cost-effectiveness analysis. Hepatology. 2017 Apr;65(4):1156-1164. doi: 10.1002/hep.28958. Epub 2017 Feb 21. PMID 27880977
- [Background] Lassailly G, Caiazzo R, Buob D, Pigeyre M, Verkindt H, Labreuche J, Raverdy V, Leteurtre E, Dharancy S, Louvet A, Romon M, Duhamel A, Pattou F, Mathurin P. Bariatric Surgery Reduces Features of Nonalcoholic Steatohepatitis in Morbidly Obese Patients. Gastroenterology. 2015 Aug;149(2):379-88; quiz e15-6. doi: 10.1053/j.gastro.2015.04.014. Epub 2015 Apr 25. PMID 25917783
- [Background] Ferrannini E, Mingrone G. Impact of different bariatric surgical procedures on insulin action and beta-cell function in type 2 diabetes. Diabetes Care. 2009 Mar;32(3):514-20. doi: 10.2337/dc08-1762. No abstract available. PMID 19246589
- [Background] Klein S, Fabbrini E, Patterson BW, Polonsky KS, Schiavon CA, Correa JL, Salles JE, Wajchenberg BL, Cohen R. Moderate effect of duodenal-jejunal bypass surgery on glucose homeostasis in patients with type 2 diabetes. Obesity (Silver Spring). 2012 Jun;20(6):1266-72. doi: 10.1038/oby.2011.377. Epub 2012 Jan 19. PMID 22262157
- [Background] Rubino F, Marescaux J. Effect of duodenal-jejunal exclusion in a non-obese animal model of type 2 diabetes: a new perspective for an old disease. Ann Surg. 2004 Jan;239(1):1-11. doi: 10.1097/01.sla.0000102989.54824.fc. PMID 14685093
- [Background] Rubino F, Forgione A, Cummings DE, Vix M, Gnuli D, Mingrone G, Castagneto M, Marescaux J. The mechanism of diabetes control after gastrointestinal bypass surgery reveals a role of the proximal small intestine in the pathophysiology of type 2 diabetes. Ann Surg. 2006 Nov;244(5):741-9. doi: 10.1097/01.sla.0000224726.61448.1b. PMID 17060767
- [Background] Verdam FJ, Greve JW, Roosta S, van Eijk H, Bouvy N, Buurman WA, Rensen SS. Small intestinal alterations in severely obese hyperglycemic subjects. J Clin Endocrinol Metab. 2011 Feb;96(2):E379-83. doi: 10.1210/jc.2010-1333. Epub 2010 Nov 17. PMID 21084402
- [Background] Gniuli D, Calcagno A, Dalla Libera L, Calvani R, Leccesi L, Caristo ME, Vettor R, Castagneto M, Ghirlanda G, Mingrone G. High-fat feeding stimulates endocrine, glucose-dependent insulinotropic polypeptide (GIP)-expressing cell hyperplasia in the duodenum of Wistar rats. Diabetologia. 2010 Oct;53(10):2233-40. doi: 10.1007/s00125-010-1830-9. Epub 2010 Jun 30. PMID 20585935
- [Background] Rajagopalan H, Cherrington AD, Thompson CC, Kaplan LM, Rubino F, Mingrone G, Becerra P, Rodriguez P, Vignolo P, Caplan J, Rodriguez L, Galvao Neto MP. Endoscopic Duodenal Mucosal Resurfacing for the Treatment of Type 2 Diabetes: 6-Month Interim Analysis From the First-in-Human Proof-of-Concept Study. Diabetes Care. 2016 Dec;39(12):2254-2261. doi: 10.2337/dc16-0383. Epub 2016 Aug 12. PMID 27519448
- [Background] Gollisch KS, Lindhorst A, Raddatz D. EndoBarrier Gastrointestinal Liner in Type 2 Diabetic Patients Improves Liver Fibrosis as Assessed by Liver Elastography. Exp Clin Endocrinol Diabetes. 2017 Feb;125(2):116-121. doi: 10.1055/s-0042-118961. Epub 2016 Dec 22. PMID 28008583